CLINICAL TRIAL: NCT07316907
Title: An Exploratory Clinical Study of the Safety and Efficacy of Allogenic CD19-Targeted Chimeric Antigen Receptor T-Cell Injection in the Treatment of Relapsed/Refractory B-Cell Hematologic Malignancies
Brief Title: A Clinical Study of Allogenic CD19-CAR-T in the Treatment of R/R B-Cell Hematologic Malignancies
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: YANRU WANG (Other)
Collaborators: Allorunning Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, YANRU WANG, Clinical Professor, Affiliated Hospital of Jiangsu University
Organization: Affiliated Hospital of Jiangsu University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EU19
Record Dates: First submitted 2025-12-09; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Hematologic Malignancies; Lymphoma
Keywords: CD19-positive; relapsed/refractory; B-cell hematologic malignancies
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- relapsed/refractory B-cell hematologic malignancies (Experimental): relapsed/refractory B-cell hematologic malignancies patients to be treated with 19UCART cells
  Interventions: Biological: 19UCART injection

INTERVENTIONS:
Biological: 19UCART injection — 19UCART injection is a CD19-targeted allogenic CAR-T. A single infusion of CAR-T cells will be administered intravenously.

SUMMARY:
This is a single-arm, open-label pilot study to evaluate the safety and efficacy of CD19-targeted allogenic CAR-T cells (19UCART) in patients with relapsed/refractory B-cell hematologic malignancies. 12 patients are planned to be enrolled in the dose-escalation trial. The primary objective of the study is to evaluation of the safety and feasibility of 19UCART for the treatment of relapsed/refractory B-cell hematologic malignancies. The secondary objective is to evaluate the efficacy of 19UCART for the treatment of relapsed/refractory B-cell hematologic malignancies. The exploratory objective is to evaluate expansion, persistence and ability of 19UCART to deplete CD19 positive cells in patients with relapsed/refractory B-cell hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in this trial with signed informed consent.
2. Diagnosis of B-cell hematologic malignancy according to the 2017 WHO classification, including B-acute lymphoblastic leukemia (B-ALL) and mature B-cell lymphomas such as diffuse large B-cell lymphoma (DLBCL), follicular lymphoma (FL), marginal-zone lymphoma (MZL), small lymphocytic lymphoma/chronic lymphocytic leukemia (SLL/CLL), mantle-cell lymphoma (MCL), etc.
3. Refractory or relapsed B-cell malignancy defined as failure to achieve complete remission after standard therapy, or relapse after achieving remission with first-line or salvage therapy.
4. Persistence of minimal residual disease (MRD) positivity despite hematologic remission in B-cell acute lymphoblastic leukemia (ALL).
5. At least one measurable lesion ≥1.5 cm in longest diameter by IWG revised criteria for relapsed/refractory lymphoma.
6. Age 18-70 years; both sexes eligible.
7. Expected survival ≥12 weeks.
8. Adequate organ function as follows (no blood products or growth factors within 14 days before first infusion):

1). Hematology: A. White blood cell count (WBC) ≥3.0×10⁹/L B. Absolute neutrophil count (ANC) ≥1.5×10⁹/L C. Platelet count (PLT) ≥100×10⁹/L D. Hemoglobin (Hb) ≥90 g/L 2). Renal: A. Serum creatinine ≤1.5×ULN or calculated creatinine clearance ≥60 mL/min 3). Cardiac: A. Left ventricular ejection fraction (LVEF) ≥50 % B. QTc (Fridericia) ≤450 ms (men) or ≤470 ms (women) 4). Hepatic: A. Total bilirubin ≤1.5×ULN B. Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤2.5×ULN (≤5×ULN if liver involvement) 5). Coagulation: A. International normalized ratio (INR) or Prothrombin time (PT) ≤1.5×ULN B. Activated partial thromboplastin time (APTT) ≤1.5×ULN 6). Pulmonary: Diffusing capacity of the lung (DLCO) ≥50 % of predicted (with or without correction for anemia/alveolar volume).

9. ECOG performance status 0-2 at screening. 10. LVEF ≥50 % and no pericardial effusion. 11. At least 2 weeks since last prior therapy (radiation, chemotherapy, monoclonal antibody, or other systemic treatment).

12. Recovery to ≤CTCAE Grade 1 for any preceding serious adverse event (SAE). 13. WOCBP* not surgically sterilized must use highly effective contraception from study start through 6 months after last dose; men with WOCBP partners must use highly effective contraception through 3 months after last dose. WOCBP must have negative serum β-hCG within 7 days before first dose and must not be breastfeeding.

14. Ability to comply with study visit schedule and all protocol requirements.

*WOCBP = women of child-bearing potential

Exclusion Criteria:

* Subjects with any of the following conditions are ineligible for this trial:

  1. Known hypersensitivity, allergic reaction, intolerance, or contraindication to 19UCART or any study-drug component (including fludarabine, cyclophosphamide, or tocilizumab), or history of severe anaphylaxis.
  2. Post-allo-HSCT relapse with active graft-versus-host disease requiring systemic corticosteroids or other immunosuppressants.
  3. Uncontrolled active infection of any etiology.
  4. Active hepatitis B, hepatitis C, or tuberculosis.
  5. HIV or syphilis infection.
  6. Active autoimmune disease or history of severe autoimmune disorder (as judged by the PI) requiring prolonged immunosuppressive therapy.
  7. Congenital or acquired immunodeficiency syndromes.
  8. New York Heart Association (NYHA) class III or IV heart failure, unstable angina, myocardial infarction within 6 months, or sustained (>30 s) ventricular arrhythmia.
  9. History of epilepsy or other significant central nervous system disorders.
  10. Extra-nodal lymphomatous involvement of brain, lung, or gastrointestinal tract.
  11. Prior malignancy other than:

      1. Curatively resected non-melanoma skin cancer (e.g., basal-cell carcinoma)
      2. Curatively treated carcinoma in situ (cervical, bladder, breast, etc.)
  12. Systemic high-dose corticosteroids within 2 weeks before study entry.
  13. Pregnancy, lactation, or intention to become pregnant within 6 months.
  14. Participation in another clinical trial within 1 month.
  15. Anticipated need for any other systemic anti-neoplastic therapy during the study.
  16. Major surgery within 14 days before first study-drug administration.
  17. Any condition that, in the investigator's opinion, could increase patient risk or interfere with study results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Toxicity and adverse-event grading after 19UCART treatment | up to 12 months after infusion
  all toxicities and AEs will be assessed according to the National Cancer Institute CTCAE v5.0
CRS grading after 19UCART treatment | up to 12 months after infusion
  CRS will be graded using the Lee DW et al. CRS grading scale

SECONDARY OUTCOMES:
Overall response rate (ORR = CR + PR) of patients receive 19UCART treatment | 1, 3, 6, and 12 months after infusion
  according to the Lugano criteria and CSCO guidelines
Disease control rate (DCR = CR + PR + SD) of patients receive 19UCART treatment | 1, 3, 6, and 12 months after infusion
  according to the Lugano criteria and CSCO guidelines
PET-CT Response Criteria according to Lugano metabolic response categories | 1, 3, 6, and 12 months after infusion
  Tumor measurements and evaluations must be performed with the same technique used at baseline. CMR (5-PS 1-3 in all baseline sites); PMR (5-PS 4-5 but uptake ↓ vs base or ΔSUVmax ↓ ≥ 25 %); NMR (5-PS 4-5 with no significant Δ); PMD (5-PS 4-5 and uptake ↑ > 50 % or new lesion). Deauville 5-Point Scale (5-PS): Scores 1-3 = metabolic CR; 4-5 = residual disease.
CAR copies and cell count of CAR-T in blood after 19UCART treatment | Day 0, 1, 3, 5, 7, 9, 11, 14, 21, 28, and month 2, 3, 6, 9, 12 after infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No